CLINICAL TRIAL: NCT01339234
Title: Body-weight Supported Treadmill Training in Primary Progressive Multiple Sclerosis: A Pilot Trial
Brief Title: Supported Treadmill Training for Progressive Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hicks, Audrey, Ph.D. (Individual)
Collaborators: Multiple Sclerosis Society of Canada (Other)
Responsible Party: Audrey Hicks, McMaster University
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: Hicks -MS treadmill
Record Dates: First submitted 2011-04-18; First posted 2011-04-20 (Estimated); Last update posted 2011-04-20 (Estimated); Status verified 2011-04

CONDITIONS: Multiple Sclerosis
Keywords: treadmill exercise; rehabilitation; progressive multiple sclerosis; functional ability; quality of life; fatigue
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Chronic Progressive; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Body-weight supported treadmill training (Experimental)
  Interventions: Other: Body-weight supported treadmill training

INTERVENTIONS:
Other: Body-weight supported treadmill training — Patients will undergo training using the Woodway Loco-system which consists of a treadmill with an overhead pulley system connected to a support harness. BWSTT allows patients with limited mobility to safely walk upright on a treadmill with a portion of their body weight counter balanced. Three trainers will be required to assist with the BWSTT program. Two trainers will be positioned at the lower limbs to manually guide the participant through a proper gait motion and provided lower limb control. A third trainer will stand behind the participant to provide trunk support and assist with weight shifting.

SUMMARY:
This study is a pilot trial to evaluate the effects of supported treadmill walking in patients with primary progressive multiple sclerosis (MS) on functional and psychosocial outcomes. Patients will exercise three times per week over the course of 6 months and will be evaluated at baseline, 12 weeks and 24 weeks into the program. Follow-up testing will also be conducted 12 weeks after participants have stopped exercising to determined the lasting effects of the intervention.

The investigators hypothesize that supported treadmill walking will be effective at improving physical physical function and psychosocial outcomes in patients with primary progressive MS.

DETAILED DESCRIPTION:
The use of exercise as an adjunct to other disease modifying treatments in MS has found increasing support over the past decade. There is ample evidence that exercise therapy can improve physical measures of disability in MS, in addition to being safe and well-tolerated. However, there is a paucity of data on whether exercise is equally effective for those with primary progressive MS as it is in relapsing remitting MS. In addition, studies of exercise therapy have traditionally excluded MS patients with severe disability. There are also currently no treatments for primary progressive MS, so finding a safe disease-modifying therapy is of the utmost importance. The investigators are therefore conducting a pilot trial to evaluate the effects of exercise in the form of supported treadmill walking for patients with primary progressive MS with severe functional impairments.

Six patients with primary progressive MS with high disability level will be recruited to participate in this study. Participants will exercise using body-weight supported treadmill training (BWSTT; Woodway Loco-system) which allows a portion of an individual's body-weight to be counterbalanced by an overhead pulley system. This system allows patients with limited mobility to walk upright on the treadmill with therapist assistance. Therapists trained in using the BWSTT system will guide the patients' legs through a proper gait motion and assist with lower limb control. Participants will complete 72 training sessions (30min/session, 3x/week) over the course of 24 weeks. Participants will be evaluated at baseline, 12 weeks (half-way through the training program) and 24 weeks (end of intervention). A follow-up assessment will also be performed 12 after participants have completed the training program (36 weeks). Outcome measures are described below.

ELIGIBILITY:
Inclusion Criteria:

* Signed, written informed consent
* Males or non-pregnant females, 18-60 years of age (inclusive)
* Clinically definite PPMS as per the diagnostic criteria of Thompson et al (2000)
* Expanded disability status score 5.0-8.0 (constant assistance required)
* Body weight <90kg (due to support limitations of treadmill)
* Approval from physician to participate in the exercise program
* Ability to tolerate upright locomotion of the body weight supported treadmill
* Ability to visit the different sites required for the study
* Ability to commit to 3 weekly training sessions for the duration of 24 weeks

Exclusion Criteria:

* Any disability acquired from trauma or another illness that could interfere with evaluation of disability due to MS
* Any other serious medical condition that might impair the subject's ability to walk on a treadmill and/or participate in aerobic exercise (including but not limited to: documented heart disease or unstable angina, uncontrolled cardiac dysrhythmia, chronic obstructive lung disease, recent non-traumatic fracture, osteoporosis and severe skin ulcerations)
* Female patients who do not agree to use effective contraceptive method(s) during the study
* Current use or use within the last 2 months of any on- or off-label disease-modifying therapy including IFN-β, glatiramer acetate, IV steroids, mitoxantrone, azathioprine, and cyclophosphamide
* Previous experience with supported treadmill training
* Kidney disease, peripheral vascular disease or poor circulation
* Inability to undergo MRI or MRI with gadolinium administration

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2008-04; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Multiple Sclerosis Functional Composite (MSFC) at 12, 24 and 36 weeks | Repeat assessments: baseline, 12 weeks, 24 weeks and 36 weeks (12 weeks post-exercise follow-up)
  The MSFC assesses functional ability with three scales: the 25ft walk (leg strength and ambulation), the 9-hole peg test (arm strength and coordination) and the Paced Auditory Serial Addition Test (PASAT; cognition). Scores on all three measures are combined to produce a composite Z-score.

SECONDARY OUTCOMES:
Change from baseline in Expanded Disability Status Scale (EDSS) at 12, 24 and 36 weeks | Repeat assessments: baseline, 12 weeks, 24 weeks and 36 weeks (12 weeks post-exercise follow-up)
  The EDSS provides a measure of physical and neurological function specifically in MS patients and is scored from 0-10. This will be assessed by a train neurologist.
Change from baseline in Modified Fatigue Impact Scale (MFIS) at 12, 24 and 36 weeks | Repeat assessments: baseline, 12 weeks, 24 weeks and 36 weeks (12 weeks post-exercise follow-up)
  The MFIS is a 21-item self-report questionnaire that evaluates fatigue overall fatigue, as well as within three categories: physical (pMFIS); cognitive (cMFIS); and psychosocial (psMFIS), over the previous 4 weeks. Scores range from 0-4 on each item with a maximum total score of 84, where higher scores indicate greater fatigue levels.
Change from baseline in Multiple Sclerosis Quality of Life-54 questionnaire at 12, 24 and 36 weeks | Repeat assessments: baseline, 12 weeks, 24 weeks and 36 weeks (12 weeks post-exercise follow-up)
  The MSQOL-54 is an MS-specific measure of quality of life that consists of 54 items divided into 12 multi-item scales, 2 single-item scales, and 2 composite scores (physical and mental health).
Change from baseline in brain-derived neurotrophic factor (BDNF) at 12, 24 and 36 weeks | Repeat assessments: baseline, 12 weeks, 24 weeks and 36 weeks (12 weeks post-exercise follow-up)
Change from baseline in magnetic resonance imaging (MRI) outcomes at 24 weeks | Repeat assessments: baseline and 24 weeks
  Both standard and unconventional MRI techniques will be used to evaluate the effects of exercise on brain health.

CONTACTS AND LOCATIONS:
Overall Officials: Michel Rathbone, MD, PhD, Principal Investigator — McMaster University; Audrey Hicks, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University (Centre for Health Promotion and Rehabilitation)/Hamilton Health Sciences, Hamilton, Ontario, Canada

REFERENCES:
- [Result] Pilutti LA, Lelli DA, Paulseth JE, Crome M, Jiang S, Rathbone MP, Hicks AL. Effects of 12 weeks of supported treadmill training on functional ability and quality of life in progressive multiple sclerosis: a pilot study. Arch Phys Med Rehabil. 2011 Jan;92(1):31-6. doi: 10.1016/j.apmr.2010.08.027. PMID 21187202